CLINICAL TRIAL: NCT07197684
Title: Effect of Ultrasound Guided Pecs Block With Intravenous Ketamine and Ketamine Infusion Alone For Prevention of Chronic Post-Surgical Pain in Patients Undergoing Breast Cancer Surgery: A Randomized Controlled Trial
Brief Title: Ultrasound Guided Pecs Block and Ketamine Infusion for Preventing Chronic Pain in Patients Undergoing Breast Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ali Sarfraz Siddiqui, Assistant professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-11608-35490
Record Dates: First submitted 2025-08-29; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Pain, Chronic; Post Surgical Pain
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Pain, Postoperative | interventions — Ketamine; Nalbuphine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group K (Experimental): Intravenous Nalbuphine 0.1 mg/kg Paracetamol 1g or 15mg/kg (if weight is < 50kg).
  Additionally, before skin incision, a bolus 0.35 mg/kg ketamine will be given followed by a continuous infusion 0.25 mg/kg/hr (11) will be administered. Ketamine infusion will be stopped 30 minutes before the end of the surgery.
  Interventions: Drug: Ketamine; Drug: Nalbuphine; Drug: Paracetamol
- Group K+ Pecs (Experimental): Intravenous Nalbuphine 0.1 mg/kg Paracetamol 1g or 15mg/kg (if weight is < 50kg).
  Additionally, before skin incision, a bolus 0.35 mg/kg ketamine will be given followed by a continuous infusion 0.25 mg/kg/hr (11) will be administered. Ketamine infusion will be stopped 30 minutes before the end of the surgery.
  Additionally, Pecs block will be performed before surgical incision with the help of an ultrasound (US) by experienced anesthesiologist. The drug used for the pecs block will be two syringes of 10ml and 20 ml containing bupivacaine 0.25% (total 30 ml).
  Interventions: Drug: Ketamine; Procedure: Pecs block; Drug: Nalbuphine; Drug: Paracetamol
- Group C (Active Comparator): Intravenous Nalbuphine 0.1 mg/kg Paracetamol 1g or 15mg/kg (if weight is < 50kg).
  Interventions: Drug: Nalbuphine; Drug: Paracetamol

INTERVENTIONS:
Drug: Ketamine — Before skin incision, a bolus 0.35 mg/kg ketamine will be given followed by a continuous infusion 0.25 mg/kg/hr.
  Ketamine infusion will be stopped 30 minutes before the end of the surgery
  Arms: Group K; Group K+ Pecs
Procedure: Pecs block — Pecs block will be performed before surgical incision with the help of an ultrasound (US) by experienced anesthesiologist. The drug used for the pecs block will be two syringes of 10ml and 20 ml containing bupivacaine 0.25% (total 30 ml).
  Arms: Group K+ Pecs
Drug: Nalbuphine — Intravenous Nalbuphine 0.1 mg/kg
Drug: Paracetamol — Intravenous Paracetamol 1g or 15mg/kg (if weight is < 50kg).

SUMMARY:
The goal of this clinical trial is to is to compare the effectiveness of ultrasound-guided Pecs block with intravenous ketamine versus intravenous ketamine infusion alone in preventing Chronic Post-Surgical Pain (CPSP) in patients undergoing breast cancer surgery. The main question it aims to answer is,

How effective is the ketamine and ketamine with pecs block in reducing the frequency of Chronic Post-Surgical Pain after breast cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients with breast cancer aged between 18-75 years
* ASA (American Society of Anesthesia) physical status I, II, and III
* Patients scheduled for elective breast cancer surgery (Mastectomy with or without axillary clearance)

Exclusion Criteria:

* Refusal to participate or withdrawal of informed consent
* Surgical procedures involving breast reconstruction with flaps or implants
* Patient scheduled for bilateral mastectomy
* Reoperation on the same side due to cancer recurrence
* Known allergy or contraindication to study drugs
* History of severe psychiatric illness (e.g., major depression, bipolar disorder, schizophrenia)
* Chronic opioid use, substance abuse, or opioid addiction
* Pre-existing chronic pain or neuropathic pain disorders
* Coagulopathy, anticoagulation therapy, or localized infection at the site of block
* Uncontrolled hypertension and ischemic heart disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of Chronic Post-operative Pain | Data will be collected from patients in the breast clinic or via telephone at one week, 1,2, 3, and 6 months after surgery.
  Pain intensity will be assessed using an 11-point numeric rating scale (NRS) by an investigator blinded to group allocation. Scores range from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating greater pain severity and therefore a worse outcome.
  Data will be collected from patients in the breast clinic or via telephone at one week, 1,2, 3, and 6 months after surgery.
  All patients will be followed till six months after discharge from the hospital.

SECONDARY OUTCOMES:
Character of Chronic Post-Surgical Pain | Till six months after discharge from the hospital.
  Patients will be asked to describe the character(quality) of their pain (e.g., burning, sharp, pricking, electric-shock-like) during follow-up visits.
  patients will be subjectively asked to describe the quality of pain.
Duration of Chronic Post-Surgical Pain | Till six months after discharge from the hospital.
  From three months to six months.
Distribution of Chronic Post-Surgical Pain | Till six months after discharge from the hospital.
  Patients will be asked to report the location of any persistent pain during follow-up visits. Using a standardized body map diagram, they will indicate whether pain is present at the surgical site or in surrounding areas (e.g., axilla, upper arm, upper back, chest wall).

IPD SHARING:
Plan to Share IPD: No